CLINICAL TRIAL: NCT03591614
Title: A Pilot Study of Dendritic Cell DKK1 Vaccine for Patients With Monoclonal Gammopathy and Stable or Smoldering Myeloma
Brief Title: Dendritic Cell DKK1 Vaccine for Monoclonal Gammopathy and Stable or Smoldering Myeloma
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: PI left institution
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE1A16
Record Dates: First submitted 2018-07-09; First posted 2018-07-19 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Monoclonal Gammopathy; Smoldering Myeloma; Myeloma
Keywords: Vaccine; DKK1
MeSH Terms: conditions — Paraproteinemias; Smoldering Multiple Myeloma; Neoplasms, Plasma Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dendritic cell DKK1 vaccine (Experimental): 5-10x106 DKK1 loaded dendritic cells. Three doses will be given two weeks apart, followed by 11 months of observations.
  Interventions: Biological: DKK1

INTERVENTIONS:
Biological: DKK1 — The investigational agent is a DKK1 peptide-loaded autologous dendritic cell vaccine dispensed at a dose of 5-10x106 in 0.5 mL Plasma-Lyte A + 5% HSA.

SUMMARY:
The purpose of this study is to study the safety and preliminary efficacy of a dendritic cell DKK1 vaccine against myeloma. Dendritic cells are immune cells that are collected from the blood of the patient at Case Western Reserve Medical Center and then brought into contact with DKK1, a molecule that is present of myeloma cells but not to a significant amount on other cells except for the prostate and the placenta. It is an investigational (experimental) vaccine that based on studies in the laboratory and in mice is expected to work by presentation of DKK1 to anticancer immune cells via dendritic cells leading to an immune attack on myeloma cells. It is experimental because it is not approved by the Food and Drug Administration (FDA).

DETAILED DESCRIPTION:
The overall objective of this pilot study is to determine the safety and preliminary efficacy of a dendritic cell DKK1 vaccine in view of possible future use as a strategy to prevent progression of asymptomatic plasma cell disorders, maintain disease control, and ultimately contribute to eradication of multiple myeloma, light and heavy chain amyloidosis, immunoglobulin deposition disease, and other malignant and non-malignant diseases related to transformed plasma cells.

Primary Objective Confirm the safety of dendritic cell DKK1 vaccine given every two weeks for three doses in patients with monoclonal gammopathy, stable or smoldering myeloma.

Secondary Objectives

1. Assess response according to international response criteria (> partial response, PR) and clinical benefit response (>minor response, MR, according to adapted EBMT criteria)
2. Determine time to progression
3. Describe progression-free and overall survival

Correlative Objectives

1. Explore correlation between myeloma DKK1 and PDL-1 expression and response
2. Determine cellular immune response
3. Assess serologic anti-DKK1 antibody response

Study design including dose escalation / cohorts Pilot study with 3 patient safety run-in, possible dose level -1 (DL-1) if dose limiting toxicity occurs in one or more patients at the target dose level, and, at the first dose level where no dose limiting toxicity occurs, extension by 12 patients.

DLT will be defined as any vaccine related toxicity > grade 3 that does not resolve to grade < 2 within 7 days. If any DLT occurs at DL-1 enrollment will be stopped and an amendment will be discussed.

ELIGIBILITY:
Inclusion Criteria:

* At any time prior to enrollment subjects must have IgG, IgA, kappa, or lambda monoclonal gammopathy confirmed in at least two assessments at least three months apart or histologically confirmed multiple myeloma or carry a diagnosis of smoldering myeloma based on prior documentation of serum m-spike (IgG or IgA) of at least 3g/dL serum m-spike (IgG or IgA) or 24h urine m-spike of at least 500mg/24h.
* Within 28 days prior to enrollment persistence of the clonal plasma cell disorder must be documented by presence of a clonal band on immunofixation of blood or urine or an abnormal serum free kappa/lambda ratio.
* Subjects with myeloma related organ dysfunction must have received prior therapy, reached at least partial remission with at least one of any number of prior regimens, and be candidates for observation off myeloma therapy based on lack of progression at least stable disease for at least 90 days prior to at study entry.
* Performance status ECOG performance status ≤ 2.
* Subjects must have laboratory test results within the following ranges:

  * Hemoglobin ≥ 9.0 g/dl
  * Absolute neutrophil count ≥ 1,500/mcL
  * Platelet count ≥ 100,000/mcL
  * Total bilirubin < 2.5 x institutional upper limit of normal
  * AST (SGOT) ≤ 2.5 X institutional upper limit of normal
  * ALT (SGPT) ≤ 2.5 X institutional upper limit of normal
  * Calculated creatinine clearance (Cockcroft-Gault) ≥ 30ml/min
* Anti-myeloma treatment with proteasome inhibitors, IMiDsTM, corticosteroids, low dose cyclophosphamide (≤ 50mg per day) must have been discontinued at least 14 days prior to study entry. Conventional chemotherapy at conventional doses including cyclophosphamide at > 50mg per day must have been discontinued at least 28 days prior to study entry. At least 180 days must have passed since high dose chemotherapy used in the context of autologous stem cell transplantation. Prior radiation must have been completed at least 14 days prior to enrollment.
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Subjects receiving any other investigational agents.
* Concurrent use of any plasma cell directed therapy including corticosteroids (use of bisphosphonates is allowed).
* Subjects who have previously received an allogeneic stem cell transplant.
* Subjects with uncontrolled intercurrent illness including, but not limited to ongoing or active infection (including active HIV or hepatitis), symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Women with childbearing potential (last menstrual period within less than 24 months unless hysterectomy or bilateral oophorectomy has been performed since) as well as pregnant women are excluded from this study because DKK1 is expressed in placental tissue and a DKK1 immune response could harm the child. Breastfeeding women are excluded from this study because antibodies made in response to the dendritic cell DKK1 vaccine could enter milk and affect the health of the breastfed child.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with dose limiting toxicity | Up to 1 year
  Toxicity will be assessed according to CTCAE v.4.03. Patients will have weekly CBC w. Differential, CMP, history, and physical. DLT will be defined as any vaccine related non-hematologic toxicity, neutropenia, anemia or thrombocytopenia > grade 3 that does not resolve to grade < 2 within 7 days.

SECONDARY OUTCOMES:
Average time of progression-free survival | Up to 1 year
  Progression-free survival will be measured from administration of the first vaccine dose to progression as defined by updated uniform international response criteria or death of any cause, whichever comes first.
Average time of overall survival | Up to 1 year
  Overall survival will be measured from administration of the first vaccine dose to death from any cause.
Average time to progression | Up to 1 year
  Time to progression will be measured from administration of the first vaccine dose to progression as defined by updated uniform international response criteria
Best overall response | Up to 1 year
  Response will be evaluated according to updated uniform response criteria
Clinical Benefit Response | Up to 1 year
  Response will be evaluated according to updated uniform response criteria

CONTACTS AND LOCATIONS:
Overall Officials: Ehsan Malek, MD, Principal Investigator — University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - University Hospitals Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic, Case Comprehensive Cancer Center, Cleveland, Ohio